CLINICAL TRIAL: NCT03727347
Title: Clinical Evaluation of Low Power Radiofrequency Energy Applied to the Posterior Nasal Nerve Area for Symptomatic Relief of Chronic Rhinitis
Brief Title: Posterior Nasal Nerve (PNN) Rhinitis Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aerin Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP668
Record Dates: First submitted 2018-10-24; First posted 2018-11-01 (Actual); Results first posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2020-09

CONDITIONS: Chronic Rhinitis

STUDY DESIGN:
Intervention Model Description: All enrolled subjects will be treated with the InSeca Stylus
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- InSeca Stylus Treatment Group (Experimental): Subjects treated with low power radiofrequency energy applied to the nasal cavity mucosa overlying the region of the posterior nasal nerve (the posterior middle meatus and posterior inferior meatus)
  Interventions: Device: InSeca Stylus

INTERVENTIONS:
Device: InSeca Stylus — Low power radiofrequency energy delivery to the portion of the nasal cavity mucosa overlying the region of the posterior nasal nerve (the posterior middle meatus and posterior inferior meatus).

SUMMARY:
Evaluation of the Aerin Medical Device used for the treatment of chronic rhinitis

DETAILED DESCRIPTION:
This is a non-significant risk, prospective, multi-center, non-randomized study to evaluate the safety and efficacy of the Aerin Medical device (InSeca Stylus) when used to deliver radiofrequency (RF) energy to the posterior nasal nerve area to improve symptoms in those diagnosed with chronic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22 to 75 years (inclusively)
2. Willing and able to provide informed consent
3. Willing and able to comply with the subject-specific requirements outlined in the study protocol
4. Seeking treatment for chronic rhinitis symptoms of at least 6 months duration and willing to undergo an office-based procedure
5. Moderate to severe symptoms of rhinorrhea (rTNSS rating of 2 or 3 for rhinorrhea)
6. Mild to severe symptoms of nasal congestion (rTNSS rating of 1, 2 or 3 for congestion)
7. rTNSS score of greater than or equal to 6
8. Dissatisfaction with medical management, defined as usage of intranasal steroids for a minimum of 4 weeks without adequate symptom relief, as judged by the subject

Exclusion Criteria:

1. Anatomic obstructions that in the investigator's opinion limit access to the posterior nose
2. Altered anatomy of the posterior nose as a result of prior sinus or nasal surgery or injury
3. Active nasal or sinus infection
4. Moderate to severe ocular allergic symptoms (such as eye tearing [epiphora], itching [pruritus], or redness [erythema])
5. History of significant dry eye
6. History of any of the following: nose bleeds in the past 3 months, rhinitis medicamentosa, head or neck irradiation
7. Known or suspected allergies or contraindications to the anesthetic agents and/or antibiotic medications to be used during the study procedure session
8. Known or suspected to be pregnant, or is lactating
9. Participating in another clinical research study
10. Other medical conditions which in the opinion of the investigator would predispose the subject to poor wound healing, increased surgical risk, or poor compliance with the requirements of the study

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: V. Vasu Kakarlapudi, MD, Principal Investigator — Advanced ENT and Allergy, New Albany, IN
Locations (5):
- United States (5):
  - Colorado ENT and Allergy, Colorado Springs, Colorado
  - Advanced ENT and Allergy, New Albany, Indiana
  - Piedmont ENT Associates, Winston-Salem, North Carolina
  - Fort Worth ENT, Fort Worth, Texas
  - ENT and Allergy Associates of Texas, McKinney, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quillen DM, Feller DB. Diagnosing rhinitis: allergic vs. nonallergic. Am Fam Physician. 2006 May 1;73(9):1583-90. PMID 16719251
- [Background] Wallace DV, Dykewicz MS, Bernstein DI, Blessing-Moore J, Cox L, Khan DA, Lang DM, Nicklas RA, Oppenheimer J, Portnoy JM, Randolph CC, Schuller D, Spector SL, Tilles SA; Joint Task Force on Practice; American Academy of Allergy; Asthma & Immunology; American College of Allergy; Asthma and Immunology; Joint Council of Allergy, Asthma and Immunology. The diagnosis and management of rhinitis: an updated practice parameter. J Allergy Clin Immunol. 2008 Aug;122(2 Suppl):S1-84. doi: 10.1016/j.jaci.2008.06.003. No abstract available. PMID 18662584
- [Background] Behrbohm H. The Dual Character of Nasal Surgery. In: Behrbohm H, Tardy MEJ, eds. Essentials of Septorhinoplasty. Stuttgart, Germany: Thieme; 2004
- [Background] Geurkink N. Nasal anatomy, physiology, and function. J Allergy Clin Immunol. 1983 Aug;72(2):123-8. doi: 10.1016/0091-6749(83)90518-3. PMID 6350406
- [Background] Dahl R, Mygind N. Anatomy, physiology and function of the nasal cavities in health and disease. Adv Drug Deliv Rev. 1998 Jan 5;29(1-2):3-12. doi: 10.1016/s0169-409x(97)00058-6. PMID 10837577
- [Background] Rogers DF. Airway goblet cells: responsive and adaptable front-line defenders. Eur Respir J. 1994 Sep;7(9):1690-706. PMID 7995400
- [Background] Schroer B, Pien LC. Nonallergic rhinitis: common problem, chronic symptoms. Cleve Clin J Med. 2012 Apr;79(4):285-93. doi: 10.3949/ccjm.79a11099. PMID 22473729
- [Background] Greiner AN, Meltzer EO. Overview of the treatment of allergic rhinitis and nonallergic rhinopathy. Proc Am Thorac Soc. 2011 Mar;8(1):121-31. doi: 10.1513/pats.201004-033RN. PMID 21364230
- [Background] Halderman A, Sindwani R. Surgical management of vasomotor rhinitis: a systematic review. Am J Rhinol Allergy. 2015 Mar-Apr;29(2):128-34. doi: 10.2500/ajra.2015.29.4141. PMID 25785754
- [Background] Kirtane MV, Rajaram D, Merchant SN. Transnasal approach to the vidian nerve: anatomical considerations. J Postgrad Med. 1984 Oct;30(4):210-3. No abstract available. PMID 6527306

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients in the specialist's clinic seeking treatment for chronic rhinitis symptoms of at least 6 months duration were approached for possible participation. Following completion of the informed consent process, baseline evaluation was conducted.
Pre-assignment Details: Three potential subjects failed to meet one or more of the inclusion/exclusion criteria.
Groups:
- InSeca Stylus: Low power radiofrequency treatment of the nasal cavity mucosa overlying the region of the posterior nasal nerve (the posterior middle meatus and posterior inferior meatus)
Period: Overall Study
Arm/Group | InSeca Stylus
Started | 50
2-week Evaluation | 50
4-week Evaluation | 50
12-week Primary Endpoint Evaluation | 50
26-week Evaluation | 48
52-week Evaluation | 47
Completed | 47
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | InSeca Stylus Treatment Group
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 29.8 (6.4)
rTNSS [Mean (Standard Deviation); unit: score on a scale] — The TNSS is an instrument used to collect patient self-rated severity of 4 nasal symptoms: rhinorrhea, nasal congestion, nasal itching, and sneezing. Each of the 4 nasal symptoms is rated on a 4-point scale with 0 = no symptoms,1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms. The maximum TNSS is 12 and indicates the most severe symptoms. The "r" in rTNSS indicates a reflective evaluation; in this study, the subject was asked to evaluate symptoms over the preceding 12 hours.
  score on a scale | 8.5 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Reflective Total Nasal Symptom Score (rTNSS)
Description: Mean change in Reflective Total Nasal Symptoms Score (rTNSS) from baseline to 12 weeks post-study procedure. Improvement (12 week score - baseline score) is signified by a negative value.
  The Reflective Total Nasal Symptom Score (rTNSS) is a patient self reported questionnaire of four nasal symptoms: rhinitis, nasal congestion, nasal itching and sneezing. Patients will report their symptoms reflected or felt over the last 12 hours. Total scores can range from 0 to 12. A higher score indicates increased symptom severity. This study will measure the mean change in the rTNSS total score from Baseline to 12 week follow up visit
Time Frame: Comparison of scores at Baseline and 12 weeks post procedure
Population: The analyzed population excludes one subject who did not complete the rTNSS questionnaire at the 12 week follow-up visit due to oversight.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | InSeca Stylus Treatment Group
Number analyzed (Participants) | 49
units on a scale | -5.1 (2.6)
Statistical Analysis 1: Comparison: InSeca Stylus Treatment Group; Test type: Superiority; p < 0.0001, t-test, 2 sided; Hypothesis was that the improvement (decrease) in rTNSS mean score, from baseline to 12 weeks, would exceed 1 point

2. Primary Outcome: Percentage of Participants With Treatment Related Adverse Events (Safety)
Description: Characterization of the type and frequency of treatment-related adverse events reported during or following the study procedure. Subjects were asked about possible side effects or adverse experiences related to the study procedure at each follow up visit. Each event was documented and identified as to its relationship and level of relatedness to the study device and/or study procedure.
  This measure includes any subject who experienced at least one event considered definitely, probably, or possibly related to the device or procedure.
Time Frame: At or following the study procedure, and up to the final study visit at 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | InSeca Stylus Treatment Group
Number analyzed (Participants) | 50
Participants | 8

3. Other Pre Specified Outcome: rTNSS Responder Rate
Description: The Reflective Total Nasal Symptom Score (rTNSS) is a patient self reported questionnaire of four nasal symptoms: rhinitis, nasal congestion, nasal itching and sneezing. Patients report their symptoms reflected or felt over the last 12 hours. Total scores can range from 0 to 12. A higher score indicates increased symptom severity.
  Subjects who showed at least a 1 point improvement (decrease) in the reflective Total Nasal Symptom Score (rTNSS) were categorized as responders. An overall responder rate of at least 55% was expected.
Time Frame: Comparison of scores at Baseline and 12 weeks post procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | InSeca Stylus Treatment Group
Number analyzed (Participants) | 49
Participants | 46

4. Other Pre Specified Outcome: Change in rTNSS Over Time
Description: Reflective Total Nasal Symptom Score (rTNSS) is a patient self reported questionnaire of four nasal symptoms: rhinitis, nasal congestion, nasal itching and sneezing. Patients report their symptoms reflected or felt over the last 12 hours. Total scores range from 0 to 12. A higher score indicates increased symptom severity.
  The mean change in the rTNSS total score from Baseline to each follow up visit: 2 weeks, 4 weeks, 12 weeks, 26 weeks and 52 weeks post procedure will be recorded.
Time Frame: Baseline to each Follow Up Visit at 2 weeks, 4 weeks, 12 weeks, 26 weeks and 52 weeks post procedure.
Population: 50 subjects were enrolled. 2 week evaluation: 1 subject missed it due to unrelated illness. 4 week evaluation: 1 subject missed it due to travel; 1 other attended the visit but did not complete the questionnaire. 12 week evaluation: All subjects attended but 1 subject did not complete the questionnaire. 26 week evaluation: 2 subjects withdrew from the study prior to the visit. 52 week evaluation: 1 additional subject was lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Treatment Group - Baseline: Data collected at baseline from enrolled participants
- Treatment Group - 2 Week Data: Data collected at 2 weeks post-study procedure
- Treatment Group - 4 Week Data: Data collected at 4 weeks post-study procedure
- Treatment Group - 12 Week Data: Data collected at 12 weeks post-study procedure
- Treatment Group - 26 Week Data: Data collected at 26 weeks post-study procedure
- Treatment Group - 52 Week Data: Data collected at 52 weeks post-study procedure
Arm/Group | Treatment Group - Baseline | Treatment Group - 2 Week Data | Treatment Group - 4 Week Data | Treatment Group - 12 Week Data | Treatment Group - 26 Week Data | Treatment Group - 52 Week Data
Number analyzed (Participants) | 50 | 49 | 48 | 49 | 48 | 47
score on a scale | 8.5 (1.8) | 4.8 (2.4) | 3.6 (2.1) | 3.4 (2.3) | 3.3 (2.1) | 3.6 (2.3)

5. Other Pre Specified Outcome: Change in rTNSS Individual Nasal Symptom Component Scores Over Time
Description: Reflective Total Nasal Symptom Score (rTNSS) is a patient self reported questionnaire of four nasal symptoms: rhinitis, nasal congestion, nasal itching and sneezing. Patients will report their symptoms reflected or felt over the last 12 hours. Total scores can range from 0 to 12. A higher score indicates increased symptom severity.
  Scores from each of the four components of the questionnaire (rhinorrhea, nasal congestion, nasal itching, and sneezing) will be evaluated at each follow up visit at 2 weeks, 4 weeks, 12 weeks, 26 weeks and 52 weeks post procedure. Individual component scores can range from 0 to 3, with a higher score indicating increased symptom severity.
Time Frame: Baseline to each Follow Up visit at 2 weeks, 4 weeks, 12 weeks, 26 weeks and 52 weeks post procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group - Baseline | Treatment Group - 2 Week Data | Treatment Group - 4 Week Data | Treatment Group - 12 Week Data | Treatment Group - 26 Week Data | Treatment Group - 52 Week Data
Number analyzed (Participants) | 50 | 49 | 48 | 49 | 48 | 47
score on a scale
  Rhinorrhea | 2.5 (0.5) | 1.6 (0.9) | 1.2 (0.8) | 1.0 (0.7) | 0.9 (0.8) | 1.1 (0.8)
  Nasal Congestion | 2.5 (0.6) | 1.5 (1.0) | 1.1 (0.8) | 1.1 (0.8) | 1.1 (0.8) | 1.2 (1.0)
  Nasal Itching | 1.7 (0.9) | 0.7 (0.8) | 0.4 (0.6) | 0.5 (0.7) | 0.5 (0.7) | 0.5 (0.7)
  Sneezing | 1.9 (0.8) | 1.0 (0.7) | 0.8 (0.6) | 0.9 (0.8) | 0.8 (0.7) | 0.8 (0.8)

6. Other Pre Specified Outcome: Response on Aerin Quality-of-Life (QOL) Assessment Items
Description: This Quality-of-Life (QOL) instrument is a 9-item patient self-reported questionnaire developed by Aerin Medical to gain understanding of the impact of chronic rhinitis on daily activities, feelings, symptoms and medication use. Each item had 5 possible answers to convey the following responses: very positive, positive, neutral, negative and very negative.
  Section 1 asks "Please indicate how often you experience the following" for 6 items. For items 1, 3, 4 and 5, those who answered "never/rarely" were considered to have a positive (favorable) response. For questions 2 and 6, those who answered "frequently/very frequently" were considered to have a positive (favorable) response. Section 2 requests "Please indicate how often you use each of the following products to help you with your chronic rhinitis". For 3 items in this section, those who answered "never/rarely" were considered to have a positive (favorable) response.
Time Frame: The QOL was to be completed by the subject at baseline prior to the treatment procedure, and at the 12 week, 26 week and 52 week visits post procedure.
Population: The baseline QOL was not completed by 4 subjects enrolled in the study. 12 week evaluation: 2 subjects failed to complete the QOL. 26 week evaluation: 2 subjects withdrew from the study prior to the 26 week visit. 52 week evaluation: 1 additional subject was lost to follow-up at this visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group - Baseline | Treatment Group - 12 Week Data | Treatment Group - 26 Week Data | Treatment Group - 52 Week Data
Number analyzed (Participants) | 46 | 48 | 48 | 47
Participants
  Section 1, Item 1: Difficulty falling asleep: Positive (favorable) response | 5 | 23 | 26 | 28
  Section 1, Item 1: Difficulty falling asleep: Neutral or Negative response | 41 | 25 | 22 | 19
  Section 1, Item 2: Good sleep throughout the night: Positive (favorable) response | 11 | 28 | 28 | 22
  Section 1, Item 2: Good sleep throughout the night: Neutral or Negative response | 35 | 20 | 20 | 25
  Section 1, Item 3: Feeling fatigued during the day: Positive (favorable) response | 3 | 17 | 14 | 14
  Section 1, Item 3: Feeling fatigued during the day: Neutral or Negative response | 43 | 31 | 34 | 33
  Section 1, Item 4: Feelings of frustration/restlessness/irritability: Positive (favorable) response | 7 | 30 | 26 | 29
  Section 1, Item 4: Feelings of frustration/restlessness/irritability: Neutral or Negative response | 39 | 18 | 22 | 18
  Section 1, Item 5: Feelings of embarrassment or self-consciousness: Positive (favorable) response | 10 | 38 | 31 | 33
  Section 1, Item 5: Feelings of embarrassment or self-consciousness: Neutral or Negative response | 36 | 10 | 17 | 14
  Section 1, Item 6: Having a good sense of overall well-being: Positive (favorable) response | 24 | 36 | 38 | 40
  Section 1, Item 6: Having a good sense of overall well-being: Neutral or Negative response | 22 | 12 | 10 | 7
  Section 2, Item 1: Oral medications: Positive (favorable) response | 10 | 20 | 17 | 19
  Section 2, Item 1: Oral medications: Neutral or Negative response | 36 | 28 | 31 | 28
  Section 2, Item 2: Nasal sprays: Positive (favorable) response | 9 | 24 | 26 | 20
  Section 2, Item 2: Nasal sprays: Neutral or Negative response | 37 | 24 | 22 | 27
  Section 2, Item 3: Nasal breathing strips: Positive (favorable) response | 41 | 45 | 46 | 45
  Section 2, Item 3: Nasal breathing strips: Neutral or Negative response | 5 | 3 | 2 | 2

ADVERSE EVENTS:
Time Frame: From study procedure through 52-week evaluation
Description: Possible adverse events related to the study procedure were assessed based on physical examinations and queries of the subjects at follow-up evaluations. Details of events were documented on a standardized case report form. Anticipated observations related to the study procedure were recorded but were not categorized as adverse events unless they required mitigation or were of greater severity, duration, or degree of incidence than anticipated.
Arm/Group | InSeca Stylus Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 2/50
Other Adverse Events (participants affected / at risk) | 31/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | InSeca Stylus Treatment Group (N=50)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — unrelated to device or procedure
acute cholecystitis (Gastrointestinal disorders) | 1 (1) — unrelated to device or procedure
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | InSeca Stylus Treatment Group (N=50)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Bronchitis (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 12 (12)
Upper respiratory tract infection/common cold (Infections and infestations) | 8 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal mucosa changes (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal bleeding (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
First publication of study results shall be made in conjunction with the results from all clinical study centers participating in the multicenter study. If results of the multi-center study have not been published in full within 18 months after completion of the study, investigator shall be free to publish results. Investigator agrees to submit all proposed publications to the sponsor at least 60 days prior submission; the company has the right to comment.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT03727347/Prot_SAP_000.pdf